CLINICAL TRIAL: NCT04801407
Title: Comparative Study Between Microvascular Decompression and Percutaneous Radiofrequency Rhizotomy for Treatment of Trigeminal Neuralgia
Brief Title: Comparative Study inTreatment of Trigeminal Neuralgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, mohmed abdelsamee ahmed, assistant lecturer neurosurgery department, Sohag University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-03-06
Record Dates: First submitted 2021-03-11; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Trigeminal Neuralgia
Keywords: trigeminal neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia

STUDY DESIGN:
Intervention Model Description: prospective case -series hospital based study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency group (Active Comparator): it is the group that will be treated with Percutaneous Radiofrequency Rhizotomy
  Interventions: Procedure: percutaneous radiofrequency trigeminal rhizotomy
- Microvascular decompression group (Active Comparator): it is the group that will be treated with Microvascular decompression
  Interventions: Procedure: Microvascular decompression of the trigeminal nerve

INTERVENTIONS:
Procedure: percutaneous radiofrequency trigeminal rhizotomy — percutaneous radiofrequency trigeminal rhizotomy is a perctaneous procedure that ablate the sensory part of the nerve and
  Arms: radiofrequency group
Procedure: Microvascular decompression of the trigeminal nerve — Microvascular decompression is a procedure that decompress the nerve from vascular conflict
  Arms: Microvascular decompression group

SUMMARY:
This study aims to evaluate the results of percutaneous radiofrequency rhizotomy and the effectiveness of microvascular decompression for the treatment of trigeminal neuralgia and Comparing between them according the different outcome parameters.

DETAILED DESCRIPTION:
This is prospective case -series hospital based study, will be conducted on 40 patients with trigeminal neuralgia treated either by percutaneous radiofrequency trigeminal rhizotomy or microvascular decompression at Sohag University Hospitals, between march 2021 and June 2022 and we will divide the the patients into two groups ,one group will be treated with percutaneous radiofrequency trigeminal rhizotomy and the other group will be treated with microvascular decompression and we will asses the results with the Barrow Neurological Institute Pain Intensity Score .

ELIGIBILITY:
Inclusion Criteria:

* Failed medical treatment more than 6 months

Exclusion Criteria:

* Coagulation disorder or hemorrhagic disease;
* Mental illness and inability to cooperate;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Barrow Neurological Institute Pain Intensity Score | 3 months
  I (no pain, no medication), II (occasional pain, not requiring medication), III (some pain, controlled with medication), IV (some pain, not controlled with medication) V (severe pain, no pain relief with medication).

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Abdelsamee Ahmed, Sohag, Sohag City, Egypt